CLINICAL TRIAL: NCT05378698
Title: Effects of Tralokinumab in the Skin: an Immunologic and Molecular Investigation (TRALIS)
Brief Title: Effects of Tralokinumab in the Skin: an Immunologic and Molecular Investigation
Acronym: TRALIS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: treatment group completed but insufficient recruitment control group
Sponsor: University of Zurich (Other)
Collaborators: Hochgebirgsklinik Davos-Wolfgang (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TRALIS/TRALO-2260
Record Dates: First submitted 2022-02-17; First posted 2022-05-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis
Keywords: Tralokinumab
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Open-randomized treatment study involving state of the art technique such as imaging mass spectrometry, classical mass spectroscopy and proteomics in patients treated with Tralokinumab during 16 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy arm (No Intervention): Healthy controls
- Tralokinumab (Active Comparator): Patients with AD
  Interventions: Drug: Application of Tralokinumab

INTERVENTIONS:
Drug: Application of Tralokinumab — 2 Arms 20 patients 5 healthy controls
  Arms: Tralokinumab

SUMMARY:
The clinical efficacy of tralokinumab has been demonstrated in the treatment of AD; its MOA however remains insufficiently understood. A better understanding of the mechanisms underlying the clinical effects of tralokinumab would be of great clinical benefit since it may ultimately help us to identify more precisely candidate patients who may benefit from a therapy with tralokinumab.

DETAILED DESCRIPTION:
Primary objective:

To detect and quantify Tralokinumab in the skin of treated AD patients and concurrently characterize the cellular and molecular changes of the cutaneous and systemic immune response

Secondary objectives:

* Clinical response analysed by SCORAD, IG, DLQI and worst daily pruritus NRS
* To identify immunologic changes on a cellular and molecular level in the skin and in the blood in correlation with Tralokinumab levels over the treatment course.
* Changes in the skin barrier function over the treatment course

Primary outcome:

Detection of Tralokinumab in lesional skin after 16 weeks of treatment in comparison to the begin of the study assessed by mass spectrometry with Parallel Reaction Monitoring (PRM) using the Orbitrap ECLIPSE mass spectrometer

Secondary outcome:

* Clinical response analysed by SCORAD, IG, DLQI and worst daily pruritus NRS
* Detection and quantification of Tralokinumab levels in skin biopsies and skin swabs using mass spectrometer-based proteomics.
* Immunologic changes on a cellular and molecular level in the skin (assessed by IMC and mass spectrometer-based proteomics) and in the blood (OLINK targeted proteomics) in correlation with Tralokinumab levels over the treatment course.
* Changes in skin impedance (as a parameter for barrier changes) measured by NeviSense
* Levels of free IL-13 in blood serum and in skin biopsies
* Levels of serum IgE (total, specific)
* Blood eosinophil counts

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria (patients):

  * Moderate to severe AD
  * EASI < 50
  * 18-65 years old
  * Subject is capable of giving informed consent
  * Signed informed consent

Inclusion criteria (Healthy controls):

* No diagnosis or history of atopic dermatitis
* 18-65 years old
* Subject is capable of giving informed consent
* Signed informed consent

Exclusion Criteria:

* Use of systemic corticosteroids or systemic immunosuppressive/immunomodulating drugs within four weeks prior to start of the study
* Use of tanning beds or phototherapy within 6 weeks prior to start of the study
* History of cancer except for treated basal cell or spinal cell carcinoma of the skin
* Active or recurrent bacterial, fungal or viral infection at the time of enrollment, including patients with evidence of Human Immunodeficiency Virus (HIV) infection, Hepatitis B and Hepatitis C infection, active or untreated latent tuberculosis.
* Female patients of childbearing potential who are pregnant or breast feeding or planning a pregnancy during the duration of the trial and/or not practicing acceptable birth control for the duration of the trial
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Concentration of Tralokinumab in lesional skin after 16 weeks of treatment | 2 years
  Concentration of Tralokinumab in lesional skin after 16 weeks of treatment in comparison to the begin of the study assessed by mass spectrometry with Parallel Reaction Monitoring (PRM) using the Orbitrap ECLIPSE mass spectrometer

SECONDARY OUTCOMES:
Clinical outcome analysed by SCORAD | 2 years
  Clinical response analysed by SCORAD (SCORing Atopic Dermatitis, 0-103, higher scores worse outcome)
Clinical outcome analysed by IGA | 2 years
  Clinical response analysed by IGA (Investigator Global Assessment, 0-4, higher scores worse outcome)
Clinical outcome analysed by DLQI | 2 years
  Clinical response analysed by DLQI (Dermatology Life Quality Index, 0-30, higher scores wose outcome
Clinical outcome analysed by worst daily pruritus NRS | 2 years
  Clinical response analysed by worst daily pruritus NRS Numerating Rating Scale, 0-10, higher values worse outcome)
Detection and quantification of Tralokinumab levels in skin biopsies | 2 years
  Detection and quantification of Tralokinumab levels in skin biopsies using mass spectrometer-based proteomics
Detection and quantification of Tralokinumab levels in skin swabs | 2 years
  Detection and quantification of Tralokinumab levels in skin swabs using mass spectrometer-based proteomics.
Immunologic changes on a cellular level in the skin | 2.5 years
  Immunologic changes on a cellular level in the skin (assessed by IMC and mass spectrometer-based proteomics) in correlation with Tralokinumab levels over the treatment course
Immunologic changes on a molecular level in the skin | 2.5 years
  Immunologic changes on molecular level in the skin (assessed by IMC and mass spectrometer-based proteomics) in correlation with Tralokinumab levels over the treatment course.
Immunologic changes on a cellular and molecular level in the blood | 2.5 years
  Immunologic changes on a cellular level in the blood (OLINK targeted proteomics) in correlation with Tralokinumab levels over the treatment course.
Immunologic changes on a molecular level in the blood | 2.5 years
  Immunologic changes on a molecular level in the blood (OLINK targeted proteomics) in correlation with Tralokinumab levels over the treatment course.
Changes in skin impendance asessed by NeviSense | 2.5 years
  Changes in skin impedance (as per parameter for barrier changes)
Levels of IL-13 in blood serum | 2.5 years
  Levels of IL-13 in blood serum
Levels of IL-13 in skin biopsies | 2.5 years
  Levels of IL-13 in skin biopsies
Blood eosinophil counts | 2 years
  Eosinophil counts in peripheral blood; normal < 0.4 g/l
Levels of total serum IgE | 2 years
  Levels of total serum IgE (kU/l)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid-Grendelmeier, Prof, MD, Principal Investigator — University of Zurich
Locations (1):
- Allergy Unit, Dept. of Dermatology, Unviersity Hosptial of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No